CLINICAL TRIAL: NCT02883933
Title: Clinical and Histological Features of Head and Neck Melanoma
Acronym: head neck-mel
Status: Completed | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: 2015Ao006
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — Data Collection

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- melanoma: Patients with melanoma.
  Interventions: Other: Data collection

INTERVENTIONS:
Other: Data collection

SUMMARY:
The worldwide incidence of cutaneous melanoma has been increasing for the last 30 years in western populations. Among all melanomas, those located on the head and neck are more frequent than expected regarding the surface of this anatomical area, occur in older subjects than melanomas at other sites and have a worse prognosis than melanomas at other sites. The question whether head and neck melanomas could be a distinct entity has been debated.

DETAILED DESCRIPTION:
Aim of the study was to compare clinical and histological characteristics between head and neck melanomas and melanomas at other sites.

ELIGIBILITY:
Inclusion Criteria:

* patients with melanoma
* melanoma diagnosed between January 2004 and December 2011
* patients living in Champagne-Ardenne

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with melanoma.
Sampling Method: Non-Probability Sample
Enrollment: 1548 (Actual)
Dates: Start 2004-01; Primary Completion 2011-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Location of melanoma | Day 0
  Location of melanoma was classified in head and neck (scalp, forehead, temples, ears, neck, eyelids, nose, cheeks and area around mouse/chin) or other location (upper limb, lower limb, trunk, hand and foot).

CONTACTS AND LOCATIONS:
Locations (1):
- Chu de Reims, Reims, France, France

REFERENCES:
- [Background] Dabouz F, Barbe C, Lesage C, Le Clainche A, Arnoult G, Hibon E, Bernard P, Grange F. Clinical and histological features of head and neck melanoma: a population-based study in France. Br J Dermatol. 2015 Mar;172(3):707-15. doi: 10.1111/bjd.13489. Epub 2015 Feb 11. PMID 25333719